CLINICAL TRIAL: NCT01782742
Title: A Double Blind Placebo Controlled Randomized Study to Evaluate the Efficacy and Safety of Bexarotene in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Bexarotene Amyloid Treatment for Alzheimer's Disease
Acronym: BEAT-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCF-IRB 12-783
Record Dates: First submitted 2013-01-29; First posted 2013-02-04 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Alzheimer's Disease
Keywords: Mild to Moderate Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Bexarotene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bexarotene treatment Arm (Active Comparator): 75 mg of Bexarotene BID for week 1, then increasing to 150 mg BID for weeks 2 to 4.
  Weeks 5 to 8 is Open-label phase (150 mg BID for 4 weeks)
  Interventions: Drug: Bexarotene
- Placebo (Placebo Comparator): 1 placebo capsule BID for week 1, then increasing to 2 placebo capsules BID for weeks 2 to 4.
  Weeks 5 to 8 is Open-label phase (150 mg BID for 4 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bexarotene — Subjects will be randomized 4:1 to receive 4 weeks of double blind treatment of either Bexarotene or Placebo
  Other Names: Targretin
  Arms: Bexarotene treatment Arm
Drug: Placebo
  Arms: Placebo

SUMMARY:
Retinoid X receptors (RXR) are nuclear receptors that have been linked to numerous metabolic pathways relevant to Alzheimer's disease (AD) and Aβ (harmful protein) production and removal. The study drug "bexarotene" is an FDA approved anti-cancer agent but is not approved for use in Alzheimer's disease. Bexarotene acts as an RXR agonist that has reduced Aβ (harmful protein) in the brain in experimental models of Alzheimer's disease.

This study aims to determine the safety and effect on abnormal proteins found in the brain (based on brain scans) of 300 mg of "bexarotene" administered for one month compared to placebo (inactive agent).

ELIGIBILITY:
Inclusion Criteria:

* Males or females 50 to 90 of age inclusive.
* Diagnosis of probable AD according to National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* Willing and able to provide informed consent by either the subject or subject's legal representative.
* Willing and able to comply with study visits, treatment plan, laboratory tests, brain imaging and other procedures.
* Subjects must have a positive 18f-AV-45 PET scan as determined by a qualified rater.
* Mini-Mental State Examinations (MMSE) score between 10-20 inclusive.
* Must have a study partner who is able and willing to comply with all required study procedures.
* Females must be postmenopausal.
* Have at least eight years of education and should have previously (in pre-AD condition) been capable of reading, writing, and communicating effectively with others in English.
* If receiving therapy with a cholinesterase inhibitor and/or memantine, the dose of these agents has been stable for at least 4 weeks prior to randomization
* Normal laboratory findings at baseline including CBC, chemistry panel, serum lipids, liver functions, TSH, and vitamin B12.
* Must consent to ApoE genotyping

Exclusion Criteria:

* Any clinically relevant neurological disorder capable of producing a dementia syndrome including Parkinson's disease, stroke, vascular dementia, dementia with Lewy bodies, frontotemporal dementia and others.
* 4 or more micro-hemorrhages (amyloid-related imaging abnormalities - hemorrhage type (ARIA-H) on baseline MRI or any evidence of amyloid-related imaging abnormalities - effusion type (ARIA-E) (Sperling et al, 2011).
* History of malignancy within the past five years with the exception of basal cell or squamous cell cancer, in-situ cervical cancer, or localized prostate cancer.
* History of seizure in the past three years prior to randomization
* Any contraindication of having brain MRI
* Any contraindication of having PET (inability to lie flat and still for the duration of the scan, intolerance to previous PET such as hypersensitivity reaction to PET ligand or imaging agent)
* The subject has any unstable medical illness including hypertension, congestive heart failure, chronic obstructive pulmonary disease, renal failure, liver failure or other organ compromise.
* Other clinically important abnormality on vital signs, physical examination, neurologic examination, laboratory results, or electrocardiogram (ECG) examination (e.g. Atrial fibrillation) that could compromise the study or be detrimental to the subject.
* The subject has received bexarotene previously.
* The subject has an allergy to bexarotene.
* Has had a PET scan in the past 12 months.
* Has had radiotherapy in the past year.
* Have participated in an investigational drug or device study within 30 days prior to Visit 2.
* Have been treated with immunomodulators to treat AD (vaccines, antibodies etc) within 6 months prior to visit 2
* Unable to swallow uncrushed oral medication in capsule form
* Have any condition or reason that, in the opinion of the investigator, which could interfere with the ability of the patients to participate or complete the trials, or places the patient at undue risk or complicates the interpretation of safety or efficacy data.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Cummings, MD, ScD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Cummings JL, Zhong K, Kinney JW, Heaney C, Moll-Tudla J, Joshi A, Pontecorvo M, Devous M, Tang A, Bena J. Double-blind, placebo-controlled, proof-of-concept trial of bexarotene Xin moderate Alzheimer's disease. Alzheimers Res Ther. 2016 Jan 29;8:4. doi: 10.1186/s13195-016-0173-2. PMID 26822146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the United States at one site. The first participant was enrolled in April 2013.
Pre-assignment Details: 49 participants were screened, 29 were screen failures, 20 participants were randomized to treatment. 1 was withdrawn after Week 4 treatment. Inclusion and exclusion criteria was the strict basis for eligibility.
Groups:
- Bexarotene Treatment Arm: 75 mg of Bexarotene BID for week 1, then increasing to 150 mg BID for weeks 2 to 4.
  Weeks 5 to 8 is Open-label phase (150 mg BID for 4 weeks)
  Bexarotene: Subjects will be randomized 4:1 to receive 4 weeks of double blind treatment of either Bexarotene or Placebo
- Placebo: 1 placebo capsule BID for week 1, then increasing to 2 placebo capsules BID for weeks 2 to 4.
  Weeks 5 to 8 is Open-label phase (150 mg BID for 4 weeks)
  Placebo
Period: Double-blind Treatment Phase
Arm/Group | Bexarotene Treatment Arm | Placebo
Started | 16 | 4
Completed | 15 | 4
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Open Label Phase
Arm/Group | Bexarotene Treatment Arm | Placebo
Started | 19 | 0
Completed | 19 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexarotene Treatment Arm | Placebo | Total
Number analyzed (Participants) | 16 | 4 | 20
Age, Customized [Mean (Standard Deviation); unit: years] — Age at Screening
  years
    Age at Screening | 74.9 (6.6) | 78.1 (8.0) | 75.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 6 | 1 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Race - Caucasian | 15 | 4 | 19
  Race - African American | 1 | 0 | 1
Years of Education [Mean (Standard Deviation); unit: years] | 14.7 (4.9) | 12.3 (3.3) | 14.2 (4.7)
Years of Cognitive Symptoms [Mean (Standard Deviation); unit: years] | 4.6 (1.9) | 2.8 (0.96) | 4.3 (1.9)
MMSE total score [Mean (Full Range); unit: units on a scale] — The MMSE evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two overlapping pentagons. A lower score indicates more cognitive impairment. The lowest score that any particular person can get is 0 and the highest score is 30.
  units on a scale | 13.7 [8 to 23] | 17.0 [11 to 23] | 14.4 [8 to 23]
ADAS-Cog score [Mean (Full Range); unit: units on a scale] — The ADAS-Cog is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. A higher score indicates more impairment. Scores from the original portion of the test range from 0 (best) to 85 (worse). A positive change indicates cognitive worsening.
  units on a scale | 49.9 [35 to 65] | 40.3 [28 to 54] | 48.0 [28 to 65]
CDR score [Mean (Full Range); unit: units on a scale] — The CDR is a clinical scale that rates the severity of dementia as absent, questionable, mild, moderate, or severe (CDR score of 0, 0.5, 1, 2, or 3, respectively). Higher score means more severe dementia rating. The score is based on interviews with the participant and study partner, using a structured interview that assesses six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care.
  units on a scale | 1.4 [0 to 2] | 1.1 [0 to 2] | 1.4 [0 to 2]
NPI score [Mean (Full Range); unit: units on a scale] — The NPI is a well validated, reliable, multi-item instrument to assess psychopathology in AD based on interview with the study partner. The NPI evaluates both the frequency and severity of 10 neuropsychiatric disturbances. Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously) as well as severity (1=mild, 2=moderate, 3=severe). The overall score and the score for each subscale are the product of severity and frequency. Overall score range from 0 meaning no disturbance to 144 meaning severe disturbance.
  units on a scale | 8.7 [0 to 29] | 7.0 [2 to 16] | 8.4 [0 to 29]
NPI Distress Score [Mean (Full Range); unit: units on a scale] — NPI distress score measures the distress that the caregiver experiences during the previous 4 weeks from the assessment date. Distress score is measured on a scale between 0 to 5. 0 being not at all distressed to 5 very severely or extremely distressed. The scores for all 12 domains are added up becomes the total score. 0 means no caregiver distress and 60 means extreme caregiver distress.
  units on a scale | 6.5 [0 to 35] | 4.3 [2 to 6] | 6.1 [0 to 35]
ADCS-ADL score [Mean (Full Range); unit: units on a scale] — The ADCS-ADL is an activities-of-daily-living inventory developed by the ADCS to assess functional performance in participants with AD (Galasko et al., 1997). Using a structured interview format, study partners are queried as to whether participants attempted each item in the inventory during the prior 4 weeks and their level of performance. Overall score range from 0 meaning fully independent to 78 meaning fully dependent on assistance for activities of daily living.
  units on a scale | 53.7 [34 to 77] | 64.5 [37 to 76] | 55.9 [34 to 77]
ApoE4 Status [Number; unit: participants]
  Non-carriers | 4 | 3 | 7
  Heterozygotes | 6 | 1 | 7
  Homozygotes | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Drug-Placebo Difference in Change From Baseline to Week 4 in the Composite Amyloid Burden of the Brain
Description: The primary study endpoint for all subjects is the change from baseline to Week 4 in amyloid burden as measured by standard uptake units regional (SUVr) on amyloid brain imaging obtained through 18F-AV-45 PET
Time Frame: Baseline to Week 4
Measure: Mean (95% Confidence Interval); unit: SUVr
Groups:
- Bexarotene: 75 mg of Bexarotene BID for week 1, then increasing to 150 mg BID for weeks 2 to 4.
  Weeks 5 to 8 is Open-label phase (150 mg BID for 4 weeks)
  Bexarotene: Subjects will be randomized 4:1 to receive 4 weeks of double blind treatment of either Bexarotene or Placebo
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 16 | 4
SUVr | -0.03 [-0.06 to 0.01] | 0.02 [-0.05 to 0.10]
Statistical Analysis 1: Comparison: Bexarotene vs Placebo; Test type: Superiority or Other; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.13 to 0.03]

2. Secondary Outcome: Change in MMSE Score in ALL Subjects From Baseline to Week 4
Description: The MMSE evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two overlapping pentagons. A lower score indicates more cognitive impairment. The lowest score that any particular person can get is 0 and the highest score is 30.
Time Frame: Baseline to Week 4
Measure: Mean (95% Confidence Interval); unit: points
Groups:
- Bexarotene: 75 mg of Bexarotene BID for week 1, then increasing to 150 mg BID for weeks 2 to 4.
  Bexarotene: Subjects will be randomized 4:1 to receive 4 weeks of double blind treatment of either Bexarotene or Placebo
- Placebo: 1 placebo capsule BID for week 1, then increasing to 2 placebo capsules BID for weeks 2 to 4.
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 16 | 4
points | 0.750 [-0.783 to 2.283] | 1.750 [-1.316 to 4.816]
Statistical Analysis 1: Comparison: Bexarotene vs Placebo; Test type: Superiority or Other; p = 0.57, t-test, 2 sided; Mean Difference (Final Values) = -1.000, 95% CI 2-sided [-4.428 to 2.428]

3. Secondary Outcome: Change in ADAS-Cog Score in ALL Subjects From Baseline to Week 4
Description: The ADAS-Cog is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. A higher score indicates more impairment. Scores from the original portion of the test range from 0 (best) to 85 (worse). A positive change indicates cognitive worsening.
Time Frame: Baseline to Week 4
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 16 | 4
points | 0.375 [-2.153 to 2.903] | -0.250 [-5.307 to 4.807]
Statistical Analysis 1: Comparison: Bexarotene vs Placebo; Test type: Superiority or Other; p = 0.83, t-test, 2 sided; Mean Difference (Final Values) = 0.625, 95% CI 2-sided [-5.029 to 6.279]

4. Secondary Outcome: Change in the Global Clinical Dementia Rating Score in ALL Subjects From Baseline to Week 4
Description: The CDR is a clinical scale that rates the severity of dementia as absent, questionable, mild, moderate, or severe (CDR score of 0, 0.5, 1, 2, or 3, respectively). Higher score means more severe dementia rating. The score is based on interviews with the participant and study partner, using a structured interview that assesses six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care.
Time Frame: Baseline to Week 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 16 | 4
units on a scale | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
Statistical Analysis 1: Comparison: Bexarotene vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.000, 95% CI 2-sided [0.000 to 0.000]

5. Secondary Outcome: Change in NPI Scores in ALL Subjects From Baseline to Week 4
Description: The NPI is a well validated, reliable, multi-item instrument to assess psychopathology in AD based on interview with the study partner. The NPI evaluates both the frequency and severity of 10 neuropsychiatric disturbances. Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously) as well as severity (1=mild, 2=moderate, 3=severe). The overall score and the score for each subscale are the product of severity and frequency. Overall score range from 0 meaning no disturbance to 144 meaning severe disturbance
Time Frame: Baseline to Week 4
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 16 | 4
points | -2.625 [-6.783 to 1.533] | -2.250 [-10.570 to 6.067]
Statistical Analysis 1: Comparison: Bexarotene vs Placebo; Test type: Superiority or Other; p = 0.94, t-test, 2 sided; Mean Difference (Final Values) = -0.375, 95% CI 2-sided [-9.674 to 8.924]

6. Secondary Outcome: Change in the Activities of Daily Living (ADCS-ADL) Score in ALL Subjects From Baseline to Week 4
Description: The ADCS-ADL is an activities-of-daily-living inventory developed by the ADCS to assess functional performance in participants with AD (Galasko et al., 1997). Using a structured interview format, study partners are queried as to whether participants attempted each item in the inventory during the prior 4 weeks and their level of performance. Overall score range from 0 meaning fully independent to 78 meaning fully dependent on assistance for activities of daily living
Time Frame: Baseline to Week 4
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 16 | 4
points | -1.938 [-4.861 to 0.986] | -6.500 [-12.350 to -0.653]
Statistical Analysis 1: Comparison: Bexarotene vs Placebo; Test type: Superiority or Other; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 4.563, 95% CI 2-sided [-1.975 to 11.100]

7. Primary Outcome: Primary Outcome by Genotype (ALL SUBJECTS)
Description: This measures the change from baseline on treatment compared to placebo at week 4 on composite and regional beta amyloid burden according to ApoE genotype (E-4 carriers compared to E-4 non-carriers)
Time Frame: Baseline to Week 4
Population: Change om composite and regional Beta Amyloid burden according to ApoE genotype on ALL SUBJECTS
Measure: Mean (95% Confidence Interval); unit: SUVr
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 16 | 4
SUVr
  Frontal Medial Orbital | -0.043 [-0.081 to -0.006] | -0.021 [-0.096 to 0.054]
  Anterior Cingulate | -0.040 [-0.080 to 0.000] | 0.018 [-0.061 to 0.098]
  Parietal | -0.003 [-0.034 to 0.027] | 0.044 [-0.018 to 0.105]
  Posterior Cingulate | -0.017 [-0.065 to 0.031] | 0.044 [-0.052 to 0.141]
  Precuneus | -0.027 [-0.069 to 0.014] | 0.040 [-0.043 to 0.122]
  Temporal | -0.038 [-0.075 to 0.000] | 0.016 [-0.059 to 0.090]

8. Primary Outcome: Primary Outcome by Genotype (NON ApoE4 CARRIERS)
Description: Measures changes from baseline on treatment compared to placebo at week 4 on composite and regional Beta Amyloid burden according to ApoE genotype (NON ApoE4 CARRIERS)
Time Frame: Baseline to Week 4
Population: Change in composite and regional Beta Amyloid Burden on non-ApoE4 carriers
Measure: Mean (95% Confidence Interval); unit: SUVr
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 4 | 3
SUVr
  Composite | -0.097 [-0.155 to -0.040] | 0.047 [-0.019 to 0.114]
  Frontal Medial Orbital | -0.076 [-0.146 to -0.007] | 0.005 [-0.075 to 0.085]
  Anterior Cingulate | -0.096 [-0.166 to -0.026] | 0.048 [-0.034 to 0.129]
  Parietal | -0.068 [-0.107 to -0.029] | 0.065 [0.020 to 0.110]
  Posterior Cingulate | -0.113 [-0.180 to -0.046] | 0.074 [-0.004 to 0.151]
  Precuneus | -0.127 [-0.188 to -0.066] | 0.062 [-0.008 to 0.132]
  Temporal | -0.104 [-0.162 to -0.045] | 0.031 [-0.037 to 0.098]

9. Primary Outcome: Primary Outcome by Genotype (ApoE4 CARRIERS)
Description: This measures the change from baseline on treatment compared to placebo at week 4 on composite and regional beta amyloid burden according to ApoE genotype (E-4 carriers)
Time Frame: Baseline to Week 4
Population: Change in composite and regional Beta Amyloid burden on ApoE4 carriers
Measure: Mean (95% Confidence Interval); unit: SUVr
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 12 | 1
SUVr
  Composite | -0.005 [-0.041 to 0.031] | -0.048 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Frontal Medial Orbital | -0.033 [-0.074 to 0.009] | -0.099 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Anterior Cingulate | -0.022 [-0.062 to 0.019] | -0.069 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Parietal | 0.018 [-0.013 to 0.050] | -0.019 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Posterior Cingulate | 0.015 [-0.035 to 0.065] | -0.044 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Precuneus | 0.006 [-0.031 to 0.043] | -0.027 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Temporal | -0.015 [-0.055 to 0.024] | -0.030 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively

10. Primary Outcome: Primary Outcome by Genotype (HETEROZYGOTE ApoE4 CARRIERS)
Description: This measures the change from baseline on treatment compared to placebo at week 4 on composite and regional beta amyloid burden according to ApoE genotype (HETEROZYGOTE ApoE4 CARRIERS)
Time Frame: Baseline to Week 4
Population: Change in composite and regional Beta Amyloid burden on Heterozygote ApoE4 carriers
Measure: Mean (95% Confidence Interval); unit: SUVr
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 6 | 1
SUVr
  Composite | -0.015 [-0.037 to 0.008] | -0.048 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Frontal Medial Orbital | -0.061 [-0.090 to -0.033] | -0.099 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Anterior Cingulate | -0.048 [-0.080 to -0.016] | -0.069 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Parietal | 0.034 [0.009 to 0.058] | -0.019 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Posterior Cingulate | -0.007 [-0.035 to 0.022] | -0.044 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Precuneus | 0.005 [-0.021 to 0.032] | -0.027 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively
  Temporal | -0.010 [-0.041 to 0.020] | -0.030 [NA to NA] — With 1 placebo patient, variability within the group cannot measured effectively

11. Primary Outcome: Primary Outcome by Genotype (HOMOZYGOTE ApoE4 CARRIERS)
Description: This measures the change from baseline on treatment compared to placebo at week 4 on composite and regional beta amyloid burden according to ApoE genotype (HOMOZYGOTE ApoE4 CARRIERS)
  There are no homozygote ApoE4 carriers on the placebo arm, therefore no data can be presented on this arm.
Time Frame: Baseline to Week 4
Population: Change in composite and regional Beta Amyloid burden on Homozygote ApoE4 carriers.
  There are no homozygote ApoE4 carriers on the placebo arm, therefore no data can be presented on this arm.
Measure: Mean (95% Confidence Interval); unit: SUVr
Arm/Group | Bexarotene
Number analyzed (Participants) | 6
SUVr
  Composite | 0.005 [-0.066 to 0.075]
  Frontal Medial Orbital | -0.004 [-0.077 to 0.069]
  Anterior Cingulate | 0.005 [-0.067 to 0.077]
  Parietal | 0.003 [-0.054 to 0.060]
  Posterior Cingulate | 0.037 [-0.059 to 0.133]
  Precuneus | 0.006 [-0.065 to 0.077]
  Temporal | -0.020 [-0.096 to 0.055]

12. Secondary Outcome: Secondary Outcome Measuring Serum Biomarker Outcome Level Changes From Baseline to Week 4 in Beta amyloid1-40 and Beta amyloid1-42 (ALL SUBJECTS)
Description: Change from baseline to week 4 in beta amyloid1-40 and beta amyloid1-42 serum levels comprised in secondary biomarker outcomes
Time Frame: Baseline to Week 4
Population: Change from baseline to week 4 in beta amyloid1-40 and beta amyloid1-42 serum levels comprised in secondary biomarker outcomes in ALL SUBJECTS. There were only a total of 17 subjects who were able to provide adequate blood sample for this serum biomarker analysis. Attempts for blood sample procurement for the other 3 subjects were unsuccessful.
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 13 | 4
pmol/L
  Beta Amyloid 40 | 7.186 [-3.673 to 18.045] | -5.330 [-24.910 to 14.246]
  Beta Amyloid 42 | 0.585 [-0.044 to 1.213] | -0.900 [-2.033 to 0.233]

13. Secondary Outcome: Serum Biomarker Outcome Level Changes From Baseline to Week 4 in Beta amyloid1-40 and Beta amyloid1-42 (Non ApoE4 Carriers)
Description: Change from baseline to week 4 in beta amyloid1-40 and beta amyloid1-42 serum levels comprised in secondary biomarker outcomes (non ApoE4 carriers)
Time Frame: Baseline to Week 4
Population: Change from baseline to week 4 in beta amyloid1-40 and beta amyloid1-42 serum levels in non ApoE4 carriers. Of the 7 total subjects who were non-ApoE carriers, only 6 subjects were able to provide adequate blood sample for this serum biomarker analysis. Attempts for blood sample procurement for the other 1 subject were unsuccessful.
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 3 | 3
pmol/L
  Beta Amyloid 40 | -3.503 [-22.840 to 15.836] | -8.550 [-27.890 to 10.789]
  Beta Amyloid 42 | 0.293 [-0.873 to 1.460] | -1.127 [-2.293 to 0.040]

14. Secondary Outcome: Change in the Ratio of Beta Amyloid 42 to Beta Amyloid 40 in All Subjects
Description: This measures the change in the ratio of Beta Amyloid 42 to Beta Amyloid 40 from baseline to week 4 in all subjects
Time Frame: Baseline to Week 4
Population: There were only a total of 17 subjects who were able to provide adequate blood sample for this serum biomarker analysis. Attempts for blood sample procurement for the other 3 subjects were unsuccessful.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 13 | 4
ratio | 0.001 [-0.007 to 0.008] | -0.005 [-0.019 to 0.009]
Statistical Analysis 1: Comparison: Bexarotene vs Placebo; Test type: Superiority or Other; p = 0.46, t-test, 2 sided; Mean Difference (Final Values) = 0.006, 95% CI 2-sided [-0.010 to 0.021]

15. Secondary Outcome: Change in the Ratio of Beta Amyloid 42 to Beta Amyloid 40 in Non ApoE4 Carriers
Description: This measures the change in the ratio of Beta Amyloid 42 to Beta Amyloid 40 from baseline to week 4 in non ApoE4 Carriers
Time Frame: Baseline to Week 4
Population: Of the 7 total subjects who were non-ApoE carriers, only 6 subjects were able to provide adequate blood sample for this serum biomarker analysis. Attempts for blood sample procurement for the other 1 subject were unsuccessful.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Bexarotene | Placebo
Number analyzed (Participants) | 3 | 3
ratio | 0.005 [-0.016 to 0.026] | -0.005 [-0.026 to 0.017]
Statistical Analysis 1: Comparison: Bexarotene vs Placebo; Test type: Superiority or Other; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = 0.010, 95% CI 2-sided [-0.020 to 0.040]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the time the participants signed the informed consent forms to the Post-Treatment Follow Up Visit approximating to 4 months of time when adverse events were captured
Arm/Group | Bexarotene Treatment Arm | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/4
Other Adverse Events (participants affected / at risk) | 14/16 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexarotene Treatment Arm (N=16) | Placebo (N=4)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister on toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant had a blister on 2nd toe of left foot
Elevated triglyceride levels (Hepatobiliary disorders) | 13 (13) | 0 (0)
Elevated cholesterol level (Gastrointestinal disorders) | 6 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
Sample size of this trial is small. There was 1 participant withdrawal due to adverse event. Primary outcome measures were completed by all 20 participants as anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes